CLINICAL TRIAL: NCT05343949
Title: Promoting Activity in Chronic Obstructive Pulmonary Disease (COPD): Optimising High Intensity Interval Training and Technologies, a Pilot Study
Brief Title: High Intensity Interval Training and Technologies in COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lead coordinatior has left the site, need to find alternative lead for the study
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01022019
Record Dates: First submitted 2021-11-23; First posted 2022-04-25 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients will once screened will attend on 3 visits and will perform in a random order all of below protocols:
  A - High-intensity duration and intensity: 5 seconds Rest duration: 40 seconds Number of Repetitions: 54 Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds) B - High-intensity duration and intensity: 10 seconds Rest duration: 80 seconds Number of Repetitions: 27 Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds) C - High-intensity duration and intensity: 30 seconds Rest duration: 240 seconds Number of Repetitions: 9 Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds)
Who Masked: Participant
Masking Description: Random order of the delivery of the HIIT protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT protocol ABC (Experimental): HIIT protocol A, then HIIT protocol B, then HiIT protocol C. Patients first received HIIT A -High-intensity duration and intensity: 5 seconds, Rest duration: 40 seconds, Number of Repetitions: 54, Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds).
  After a rest of at least 2 days they received HIIT B: High-intensity duration and intensity: 10 seconds, Rest duration: 80 seconds, Number of Repetitions: 27, Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds).
  After a further rest of at least 2 days they received HIIT C-High-intensity duration and intensity: 30 seconds, Rest duration: 240 seconds, Number of Repetitions: 9 Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds).
  Interventions: Other: HIIT exercise program ABC
- HIIT protocol CAB (Experimental): HIIT protocol C, then HIIT protocol A, and lastly HIIT protocol B. Patients first received HIIT C:-High-intensity duration and intensity: 10 seconds, Rest duration: 80 seconds, Number of Repetitions: 27, Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds). After a rest of at least 2 days they received HIIT A:-High-intensity duration and intensity: 5 seconds, Rest duration: 40 seconds, Number of Repetitions: 54, Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds).
  After a further rest of at least 2 day they performed HIIT protocol B:-High-intensity duration and intensity: 10 seconds, Rest duration: 80 seconds, Number of Repetitions: 27 Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds).
  Interventions: Other: HIIT exercise program CAB
- HIIT protocol BCA (Active Comparator): HIIT protocol B, then HIIT protocol C, and lastly HIIT protocol A. Patients firstly received HIIT protocol B:-High-intensity duration and intensity: 10 seconds, Rest duration: 80 seconds, Number of Repetitions: 27, Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds).
  Following at least 2 days rest the patient will receive HIIT protocol C:-High-intensity duration and intensity: 10 seconds, Rest duration: 80 seconds, Number of Repetitions: 27, Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds). After at least another 2 days rest they will lastly receive Protocol A:-High-intensity duration and intensity: 5 seconds, Rest duration: 40 seconds, Number of Repetitions: 54, Total duration of HIIT protocol: 2,430 seconds (40 minutes, 30 seconds).
  Interventions: Other: HIIT exercise program BCA

INTERVENTIONS:
Other: HIIT exercise program ABC — Delivery of 3 different exercise programs to patients with COPD to determine which program gives least breathlessness with the same exercise benefits
  Arms: HIIT protocol ABC
Other: HIIT exercise program CAB — Delivery of 3 different exercise programs to patients with COPD to determine which program gives least breathlessness with the same exercise benefits
  Arms: HIIT protocol CAB
Other: HIIT exercise program BCA — Delivery of 3 different exercise programs to patients with COPD to determine which program gives least breathlessness with the same exercise benefits
  Arms: HIIT protocol BCA

SUMMARY:
Trials in COPD have shown that HIIT leads to the same positive outcomes as constant load training but causes less breathlessness and leg discomfort during training. However, HIIT protocols in existing trials have all been different and use relatively long interval durations (30 s) and short rests. This is sub-optimal because long interval durations lead to greater breathlessness and patients may fear that they will not fully recover during short rests, potentially decreasing adherence. A novel HIIT protocol involving very brief intervals (e.g. 10 s) with longer rests may provide the same benefits with less distress due to breathlessness.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common and disabling smoking-related lung disease that is predicted to become the 3rd leading cause of death world-wide by 2030 (WHO, 2017). The economic burden of COPD in the United Kingdom is estimated by the British Lung Foundation (BLF) to be around £48.5 billion per year - higher than all other respiratory diseases, including lung cancer. Although widespread, Hull is a COPD 'hot spot' (BLF), with prevalence and mortality rates 36% and 75% higher than the national average, respectively. COPD is characterised by symptoms of breathlessness and cough that typically progress over time.

As a consequence of these symptoms, physical activity (PA) is reduced in COPD patients, with lower levels associated with higher symptom burden, hospital admissions and mortality. Breathlessness is the most commonly reported barrier to PA in COPD, resulting in a cycle of deconditioning that ultimately leads to greater breathlessness and disability.

Pulmonary rehabilitation (PR) improves symptoms and increases exercise capacity in COPD but uptake and adherence are poor. Patients with greater breathlessness are less likely to complete PR programmes which is unsurprising given that exercise-induced breathlessness can be distressing in COPD.

One potential solution is high-intensity interval training (HIIT). HIIT involves short bursts of high-intensity exercise interspersed with periods of rest. The short duration of high-intensity exercise can reduce distressing breathlessness during exercise in COPD, mitigating the most common barrier to exercise.

As mentioned above, PR participants benefit from increased exercise capacity. However, what patients can do (exercise capacity) does not always translate into what patients do (PA) and the effect of PR on PA has been disappointing.

Interventions that aim to improve PA in COPD patients have been trialed, but the quality of evidence is low and results inconsistent. Physical inactivity is the strongest predictor of mortality in COPD patients and therefore, effective interventions that increase PA are desperately needed.

ELIGIBILITY:
Inclusion Criteria:

* Mild, Moderate and severe* COPD forced expired volume (FEV-1) ≥30 with an FEV-1/ forced vital capacity (FVC) ratio <70%) confirmed on spirometry within 6 months of recruitment.

  * Chronic breathlessness that limits exercise capacity (mMRC ≥2).
  * Using inhaled therapy for COPD including a long-acting bronchodilator agonist (LABA and/or long acting muscarinic agonist (LAMA) with or without inhaled corticosteroids (ICS).
  * Oxygen saturations ≥90% breathing room air.
  * Willing and able to undertake study procedures.
  * Has provided informed consent. * Mild and Moderate COPD patients will be recruited from the start of the study. A review of exercise session completion rates and adverse events will be performed after 10 patients have been recruited to assess the tolerability and acceptability of the different HIIT protocols prior to beginning recruitment of people with severe COPD

Exclusion Criteria:

* Significant physical or psychological comorbidity considered by the investigator likely to affect study outcomes.

  * Active cardiovascular disease or recent significant cardiovascular event (myocardial infarction within 6 months, cardiac arrhythmias including atrial fibrillation/flutter within 6 months, unstable angina within 6 months, stable angina with current symptoms).
  * Moderate or severe COPD exacerbation within 4 weeks of screening (an exacerbation requiring treatment with steroids and/or antibiotics or leading to hospitalisation).
  * Unable or unwilling to undertake exercise as set out in the study protocol

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Comparison of the Change from baseline in mean Borg Dyspnoea scale (the higher the score the worst the breathlessness) following HIIT protocols | Through study completion, on average 2 wks
  The Dyspnoea Borg scale was assessed at rest and then at the beginning and end of each high intensity interval. during and following each of the HIIT protocols lasting 40 min. the scale ranges from 0-10 with 0 being no breathlessness and 10 being maximum breathlesness

SECONDARY OUTCOMES:
Comparison of maximum Dyspnoea Borg score for each HIIT protocol (the higher the score the worse the breathlessness | through study completion, on average 2 wks
  Assessed the maximum score for Dyspnoea during high intensity training for each of the HIIT protocols with 0 being no breathlessness and 10 the maximum breathlessness.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom

REFERENCES:
- [Background] Watz H, Waschki B, Meyer T, Magnussen H. Physical activity in patients with COPD. Eur Respir J. 2009 Feb;33(2):262-72. doi: 10.1183/09031936.00024608. Epub 2008 Nov 14. PMID 19010994
- [Background] Katajisto M, Kupiainen H, Rantanen P, Lindqvist A, Kilpelainen M, Tikkanen H, Laitinen T. Physical inactivity in COPD and increased patient perception of dyspnea. Int J Chron Obstruct Pulmon Dis. 2012;7:743-55. doi: 10.2147/COPD.S35497. Epub 2012 Oct 29. PMID 23152679
- [Background] Troosters T, van der Molen T, Polkey M, Rabinovich RA, Vogiatzis I, Weisman I, Kulich K. Improving physical activity in COPD: towards a new paradigm. Respir Res. 2013 Oct 30;14(1):115. doi: 10.1186/1465-9921-14-115. PMID 24229341
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Hayton C, Clark A, Olive S, Browne P, Galey P, Knights E, Staunton L, Jones A, Coombes E, Wilson AM. Barriers to pulmonary rehabilitation: characteristics that predict patient attendance and adherence. Respir Med. 2013 Mar;107(3):401-7. doi: 10.1016/j.rmed.2012.11.016. Epub 2012 Dec 19. PMID 23261311
- [Background] Candemir İ., Kaymaz D., Ergün P. The reasons for non-adherence in pulmonary rehabilitation programs. Eurasian J. Pulmonol. 2017;19:25-29
- [Background] Robinson H, Williams V, Curtis F, Bridle C, Jones AW. Facilitators and barriers to physical activity following pulmonary rehabilitation in COPD: a systematic review of qualitative studies. NPJ Prim Care Respir Med. 2018 Jun 4;28(1):19. doi: 10.1038/s41533-018-0085-7. PMID 29867117
- [Background] Kortianou EA, Nasis IG, Spetsioti ST, Daskalakis AM, Vogiatzis I. Effectiveness of Interval Exercise Training in Patients with COPD. Cardiopulm Phys Ther J. 2010 Sep;21(3):12-9. PMID 20957074
- [Background] Coronado M, Janssens JP, de Muralt B, Terrier P, Schutz Y, Fitting JW. Walking activity measured by accelerometry during respiratory rehabilitation. J Cardiopulm Rehabil. 2003 Sep-Oct;23(5):357-64. doi: 10.1097/00008483-200309000-00006. PMID 14512781
- [Background] Mantoani LC, Rubio N, McKinstry B, MacNee W, Rabinovich RA. Interventions to modify physical activity in patients with COPD: a systematic review. Eur Respir J. 2016 Jul;48(1):69-81. doi: 10.1183/13993003.01744-2015. Epub 2016 Apr 21. PMID 27103381
- [Background] Waschki B, Kirsten A, Holz O, Muller KC, Meyer T, Watz H, Magnussen H. Physical activity is the strongest predictor of all-cause mortality in patients with COPD: a prospective cohort study. Chest. 2011 Aug;140(2):331-342. doi: 10.1378/chest.10-2521. Epub 2011 Jan 27. PMID 21273294